CLINICAL TRIAL: NCT02279446
Title: Development of a Validated Chart for Intermediate Vision Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: 263/13-10-2014
Record Dates: First submitted 2014-10-13; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Myopia; Hyperopia; Presbyopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia; Astigmatism | interventions — Restraint, Physical

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 20/20ND group: This group will have 20/20 visual acuity both in distant and near.
  Interventions: Other: Intermediate Visual acuity (IVA) assessment
- 20/20D group: This group will have 20/20 distant visual acuity and variable near visual acuity.
  Interventions: Other: Intermediate Visual acuity (IVA) assessment
- 20/20N group: This group will have 20/20 near visual acuity and variable distant visual acuity.
  Interventions: Other: Intermediate Visual acuity (IVA) assessment
- s20/20ND group: This group will have variable near and distant visual acuity (both less than 20/20)
  Interventions: Other: Intermediate Visual acuity (IVA) assessment

INTERVENTIONS:
Other: Intermediate Visual acuity (IVA) assessment — Intermediate visual acuity (IVA) will be assessed with the Intermediate Visual acuity chart which is similar to the prevalent Jaeger chart. It consists of short blocks of text in various type sizes.The computer screen is set at a specific reading distance (1 meter) and the patient is asked to read the passage with the smallest type he/she can see. According to the smallest text he/she can read, IVA is classified from IVA1 (which is considered the equivalent of 20/20 distance visual acuity) to IVA5

SUMMARY:
Development of a validated computer-based instrument (software program) for the assessment of intermediate visual acuity.

DETAILED DESCRIPTION:
Development of a validated computer-based instrument (software program) for the assessment of intermediate visual acuity (IVA). It is known that no validated method for the evaluation of IVA exists.

Primary objective of the study is to validate a specific computer-based chart (optotype) that will enable: a) comparative studies among different groups of presbyopic patients with refractive errors (ie. myopia, hyperopia, and/or astigmatism), and, b) assessment of the efficacy of surgical refractive procedures (ie. LASIK) on presbyopic patients.

Intermediate Visual acuity chart is similar to the prevalent Jaeger chart. It consists of short blocks of text in various type sizes.The computer screen is set at a specific reading distance (1 meter) and the patient is asked to read the passage with the smallest type he/she can see. According to the smallest text he/she can read, IVA is classified from IVA1 (which is considered the equivalent of 20/20 distance visual acuity) to IVA5

Validation of the computer-based IVA chart will be done by correlating the results of the IVA chart to the corresponding ones from the validated 20/20 distant and Jaeger near visual acuity charts, in a random sample of study participants with different refractive errors and different near and distant visual acuities.

ELIGIBILITY:
Inclusion Criteria:

* native Greek participants or foreigners with perfect knowledge (verbal and written) of Greek language

Exclusion Criteria:

* glaucoma or suspicion for glaucoma,
* corneal disease or suspicion for corneal disease
* fundus disease or suspicion for fundus disease
* pregnancy or nursing,
* underlying autoimmune disease
* mental or neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Intermediate Visual Acuity (IVA) | 6 months
  Number of participants that their intermediate visual acuity measured with the "intermediate visual acuity chart" will be statistically correlated with distant visual acuity (measured by 20/20 chart) and near visual acuity (measured by Jaeger chart)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Director — Assistant Professor
Locations (1):
- Eye Institute Of thrace, Alexandroupoli, Evros, Greece